CLINICAL TRIAL: NCT05630417
Title: Investigation of the Effect of Geriatric Massage Applied to the Elderly With Type 2 Diabetes on Diabetes Symptoms and Blood Parameters
Brief Title: Investigation of the Effect of Geriatric Massage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayburt University (Other)
Responsible Party: Principal Investigator, Emine APAYDIN, Lecturer, Bayburt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EAPAYDIN.TEZ-KTÜ
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Nursing Caries
Keywords: Blood parameters; Elderly; Geriatric massage; Symptom; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The research was planned as a pre test-post test randomized controlled single-center study.
Who Masked: Participant, Investigator
Masking Description: In order to keep the possibility of randomization of the elderly into groups and to minimize the possibility of their interaction with each other, the elderly who applied to Bayburt State Hospital Internal Medicine Outpatient Clinic randomly on Mondays and Wednesdays with the diagnosis of Type 2 diabetes will be included in the geriatric massage group, and the elderly who apply on Tuesday and Thursday will be included in the control group. In addition, individuals will be stratified according to age (65-74 years / 75-84 years old) while being assigned to the experimental and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Geriatric Massage Group (Experimental): The fragility of the elderly, the sensitivity of skin, muscle and bone tissue necessitate modification of massage techniques according to the individual characteristics of the elderly. Geriatric massage is a form of massage applied according to the characteristics of the elderly individual and can be applied to all body parts according to the needs of the elderly. However, since diabetic neuropathy, which is a long-term complication that is common in individuals with Type 2 diabetes and can affect all body parts, shows more symptoms in the feet, foot massage as a geriatric massage may be effective in reducing diabetes symptoms and improving blood parameters. Because of its more systemic effects, back massage was preferred.
  Interventions: Other: Feet and Back Massage
- Control Group (No Intervention): No attempt will be made by the researcher on the elderly with Type 2 diabetes in the control group. The elderly in this group will benefit from the standard care practices offered by the institution.

INTERVENTIONS:
Other: Feet and Back Massage — Foot massage: Feet are the most neglected organs of people and therefore cause many complaints. Foot massage is a massage applied to the back of the foot, toes, soles of the feet, the muscles between the thumb and little fingers, and the heel, where the muscles between the metatarsal bones are located.
  Back massage: Back massage is a non-invasive nursing intervention that can be easily applied by nurses. In back massage application; A 10-minute back massage program applied by Çınar and Eşer (2012) will be applied.
  Arms: Geriatric Massage Group

SUMMARY:
There is no study has been found to examine the effect of geriatric massage applied to the elderly with type 2 diabetes on diabetes symptoms and blood parameters. This study was planned as a pretest-posttest randomized controlled single-center study to examine the effect of geriatric massage on diabetes symptoms and blood parameters in the elderly with type 2 diabetes. 60 elderly people who type 2 diabetes who applied to the Internal Medicine Polyclinic of Bayburt State Hospital in the city center of Bayburt will the diagnosis of Type 2 diabetes will form the sample of the study. The sample will consist of two groups, the geriatric massage group and the control group. Data will be collected with the "Elderly Information Form", "Standardized Mini-Mental Test", "Diabetes Symptoms Checklist Scale", "Blood Parameters Monitoring Form". "Geriatric Massage" will be applied as an intervention. The geriatric massage group will receive 20 minutes (10 minutes on each foot) foot massage and 10 minutes back massage, two days a week for eight weeks. The control group will receive the institution's standard of care. Frequency, number, mean, Student's t test and/or Mann-Whitney U test, ANOVA and/or Kruskal-Wallis test, Chi-square test and/or Correlation and Regression Analysis will be used in the analysis of the data. As a result of this study, it is anticipated that the effects of geriatric massage on diabetes symptoms and blood parameters in the elderly with Type 2 diabetes will be determined and these effects will be included in evidence-based guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-84
* No visual or hearing impairment
* Ability to communicate verbally
* Applying to Bayburt State Hospital Internal Medicine Polyclinic
* Having a diagnosis of Type 2 diabetes for at least six months
* A score of 25 and above on the Standardized Mini Mental Test
* Agreeing to participate in the research

Exclusion Criteria:

* Having vascular disease (thrombus, phlebitis, arterial embolism, severe venous ulceration)
* Having heart failure, pacemaker and neurological disease
* Body temperature being higher than 37.5°C for more than two days, suspected or diagnosed with inflammation
* Having acute pain
* Cancer and undiagnosed malignancies, receiving chemotherapy and radiotherapy
* Presence of any scar tissue, chronic inflammatory skin diseases on the back
* Having foot amputation, fracture, infection, wound, skin disease, pathology and neuropathy related to muscles and bones

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Elderly Information Form | First day
  This form, which was created by the researchers by scanning the literature, consists of two parts. In the first part, seven questions to determine the introductory characteristics of the elderly (age, gender, marital status, place of residence, education level, occupation, smoking and alcohol use); In the second part, there are a total of 13 questions, six of which are aimed at determining the diabetes characteristics of the elderly (duration of diabetes, type of treatment, regular application of treatment, presence of other chronic diseases, attention to diet, regular exercise).
Standardized Mini Mental Test (SMMT) | will be applied on the first day. If the Standardized Mini Mental Test result is not 25 points or more, the patient will be excluded.]
  This test consists of "orientation, recording, attention, calculation, reminder, language tests and configuration" sections. Test; It is a test that can be administered by physicians, nurses and psychologists in a short time (10 minutes), outpatient conditions or at the bedside. The test was developed for the purpose of short-term cognitive assessment in the elderly, especially in the examination of delirium or dementia.Each question in the test is worth "1" point. The lowest score that can be obtained from the scale is "0" and the highest score is "30". According to the points received; 0-12 points at "severe" level, 13-22 points at "moderate" level and 23-24 points at "mild" level as "cognitive impairment"; A score between 25 and 30 is considered as "no cognitive impairment".
Diabetes Symptoms Checklist Scale | First week
  This scale was developed by Grootenhuis et al. The scale assesses the physical and psychological symptoms and perceived burden of Type 2 diabetes and its complications. The scale consisting of thirty-four items; It includes six sub-dimensions: "hyperglycemia, hypoglycemia, psychology, cardiology, ophthalmatology and neurology". Each item in the scale is numbered from 0 to 5 point. If the individual with diabetes says that he/she experiences the related symptom, that is, if he/she answers "yes", he/she chooses the level of discomfort perceived by the individual on a scale from 1 to 5 point. If the person with diabetes says that there are no symptoms, the item is evaluated as "0 point". The total score and all sub-dimension scores in the scale range from 0 to 5 point, with higher scores indicating greater symptom burden.
Blood Parameters Follow-up Form | First week
  This form was created by the researcher by scanning the literature to record and monitor the blood parameters of the elderly with diabetes. in form; There are seven values including glycosylated hemoglobin (HbA1C/%), fasting plasma glucose (APG/mg/dl), triglyceride (TG/mg/dl), high-density lipoprotein (HDL/mg/dl), low-density lipoprotein (LDL/mg/dl), creatinine mg/dl and urea mg/dl values of the elderly. These seven values are routinely requested from all patients who come to Bayburt State Hospital Internal Medicine Outpatient Clinic with the diagnosis of Type 2 diabetes and the results are recorded in the computer environment. Blood parameter results will be taken from the computer environment and recorded by the researcher.

SECONDARY OUTCOMES:
Diabetes Symptoms Checklist Scale | Forth week
  This scale was developed by Grootenhuis et al. The scale assesses the physical and psychological symptoms and perceived burden of Type 2 diabetes and its complications. The scale consisting of thirty-four items; It includes six sub-dimensions: "hyperglycemia, hypoglycemia, psychology, cardiology, ophthalmatology and neurology". Each item in the scale is numbered from 0 to 5 point. If the individual with diabetes says that he/she experiences the related symptom, that is, if he/she answers "yes", he/she chooses the level of discomfort perceived by the individual on a scale from 1 to 5 point. If the person with diabetes says that there are no symptoms, the item is evaluated as "0 point". The total score and all sub-dimension scores in the scale range from 0 to 5 point, with higher scores indicating greater symptom burden.
Diabetes Symptoms Checklist Scale | Eighth week
  This scale was developed by Grootenhuis et al. The scale assesses the physical and psychological symptoms and perceived burden of Type 2 diabetes and its complications. The scale consisting of thirty-four items; It includes six sub-dimensions: "hyperglycemia, hypoglycemia, psychology, cardiology, ophthalmatology and neurology". Each item in the scale is numbered from 0 to 5 point. If the individual with diabetes says that he/she experiences the related symptom, that is, if he/she answers "yes", he/she chooses the level of discomfort perceived by the individual on a scale from 1 to 5 point. If the person with diabetes says that there are no symptoms, the item is evaluated as "0 point". The total score and all sub-dimension scores in the scale range from 0 to 5 point, with higher scores indicating greater symptom burden.
Diabetes Symptoms Checklist Scale | Twelfth week
  This scale was developed by Grootenhuis et al. The scale assesses the physical and psychological symptoms and perceived burden of Type 2 diabetes and its complications. The scale consisting of thirty-four items; It includes six sub-dimensions: "hyperglycemia, hypoglycemia, psychology, cardiology, ophthalmatology and neurology". Each item in the scale is numbered from 0 to 5 point. If the individual with diabetes says that he/she experiences the related symptom, that is, if he/she answers "yes", he/she chooses the level of discomfort perceived by the individual on a scale from 1 to 5 point. If the person with diabetes says that there are no symptoms, the item is evaluated as "0 point". The total score and all sub-dimension scores in the scale range from 0 to 5 point, with higher scores indicating greater symptom burden.
Blood Parameters Follow-up Form | Twelfth week
  This form was created by the researcher by scanning the literature to record and monitor the blood parameters of the elderly with diabetes. in form; There are seven values including glycosylated hemoglobin (HbA1C/%), fasting plasma glucose (APG/mg/dl), triglyceride (TG/mg/dl), high-density lipoprotein (HDL/mg/dl), low-density lipoprotein (LDL/mg/dl), creatinine mg/dl and urea mg/dl values of the elderly. These seven values are routinely requested from all patients who come to Bayburt State Hospital Internal Medicine Outpatient Clinic with the diagnosis of Type 2 diabetes and the results are recorded in the computer environment. Blood parameter results will be taken from the computer environment and recorded by the researcher.

CONTACTS AND LOCATIONS:
Locations (1):
- Bayburt University, Bayburt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No